CLINICAL TRIAL: NCT06372964
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Lumateperone for the Treatment of Major Depressive Episodes (MDEs) Associated With Bipolar I or Bipolar II Disorder (Bipolar Depression) in Pediatric Patients Aged 10 to 17 Years
Brief Title: Multicenter Study of Lumateperone for the Treatment of Bipolar Depression in Pediatric Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-421
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone (Experimental): Lumateperone 42 mg for patient ages 13-17 years and Lumateperone 21 mg for patient ages 10-12 years.
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone — Lumateperone administered orally, once daily.
  Arms: Lumateperone
Drug: Placebo — Matching placebo administered orally, once daily.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study in pediatric patients who are experiencing major depressive episodes (MDEs) associated with a primary diagnosis of bipolar I or bipolar II disorder as confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL), according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5).

DETAILED DESCRIPTION:
The study will be conducted in 3 phases:

* Screening Period (up to 2 weeks) during which patient eligibility will be assessed
* Double-blind Treatment Period (6 weeks) during which all patients will be randomized to receive lumateperone or placebo in 1:1 ratio.
* Safety Follow-up Period (1 week) during which all patients will return to the clinic for a safety follow-up (SFU) visit approximately one week after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide consent as follows:

   * The Legally Authorized Representative (LAR) must provide written, informed consent.
   * The patient must provide written assent;
2. Male or female patients 10 to 17 years of age, inclusive;
3. Have a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR) primary diagnosis of bipolar I or bipolar II disorder with a current MDE without psychosis as confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL);
4. Subject has a lifetime history of at least one manic or hypomanic episode.
5. Subject's current major depressive episode is ≥ 4 weeks and less than 12 months in duration;
6. CDRS-R total score ≥ 45 with ≥ 5 on Item 11 (depressed feelings) at Screening and Baseline;
7. Young Mania Rating Scale (YMRS) score ≤ 15 (with YMRS Item 1 [elevated mood] score ≤ 2) at Screening and Baseline.

Exclusion Criteria:

1. Has a primary psychiatric diagnosis other than bipolar I or bipolar II disorder. Exception includes:

   * Attention deficit hyperactivity disorder (ADHD). If a subject is taking medications for ADHD, they must have been on a stable treatment regimen of these medication(s) for 30 days prior to screening and the treatment regimen is expected to remain stable throughout the study.
2. Intellectual disability based on Investigator opinion and DSM-5 criteria
3. Patient has been hospitalized for a bipolar manic episode within the 30 days prior to randomization;
4. Demonstrates a ≥ 25% decrease (improvement) in the CDRS-R total score between Screening and Baseline visits, or the CDRS-R is below 45 at Baseline;
5. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during his/her participation in the study or

   1. At Screening, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to Screening or, at Baseline, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 since the Screening Visit;
   2. At Screening, the patient has had 1 or more suicidal attempts within the 2 years prior to Screening; or
   3. At Screening or Baseline, scores > 3 on Item 13 (suicidal ideation) on the CDRS-R; or
   4. The patient is considered to be an imminent danger to him/herself or others.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Children's Depression Rating Scale-Revised (CDRS-R) | Week 6
  The Children's Depression Rating Scale-Revised is an observer-rated, 17-item semi-structured scale for pediatric patients. The scale comprises cognitive, somatic, affective, and psychomotor symptoms of depression. Items are rated for severity on a 7-point scale (1 to 7) for 14 items and on a 5-point scale (1 to 5) for three items. Total scores range from 7 to 113.

SECONDARY OUTCOMES:
Clinical Global Impression Scale-Severity (CGI-S) | Week 6
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Locations (48):
- United States (41):
  - Clinical Site, Dothan, Alabama
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Anaheim, California
  - Clinical Site, Redlands, California
  - Clinical Site, Sacramento, California
  - Clinical Site, San Diego, California
  - Clinical Site, West Covina, California
  - Clinical Site, Colorado Springs, Colorado
  - Clinical Site, Gainesville, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Homestead, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Gardens, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, Miami Springs, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Lawrenceville, Georgia
  - Clinical Site, Savannah, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Bloomfield Hills, Michigan
  - Clinical Site, Saint Charles, Missouri
  - Clinical Site, Lincoln, Nebraska
  - Clinical Site, Kinston, North Carolina
  - Clinical Site, Avon Lake, Ohio
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Garfield, Ohio
  - Clinical Site, Westlake, Ohio
  - Clinical Site, Oklahoma City, Oklahoma
  - Clinical Site, Austin, Texas
  - Clinical Site, Flower Mound, Texas
  - Clinical Site, Frisco, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Richmond, Texas
  - Clinical Site, Richmond, Virginia
  - Clinical Site, Bellevue, Washington
  - Clinical Site, Everett, Washington
- India (4):
  - Clinical Site, Ahmedabad
  - Clinical Site, Aurangabad
  - Clinical Site, Nashik
  - Clinical Site, Varanasi
- Serbia (3):
  - Clinical Site, Belgrade
  - Clinical Site, Niš
  - Clinical Site, Novi Sad